CLINICAL TRIAL: NCT05346250
Title: Effect of Moderate and Vigorous Exercise on Incident Diabetes in Central Obese Subjects: a 10-year Follow-up Study
Brief Title: Long-term Effect of Moderate and Vigorous Exercise on Incident Diabetes in Obese Subjects
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xiaoying Li, Professor, Shanghai Zhongshan Hospital
Other Study IDs: CCEMD011V2
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes; Obesity, Abdominal
Keywords: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity, Abdominal; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non exercise program: Subjects receive 12 month lifestyle education alone.
  Interventions: Behavioral: Non-exercise control
- Moderate intensity exercise program: Subjects receive 12 month moderate exercise.
  Interventions: Behavioral: Moderate intensity exercise
- Vigorous intensity exercise program: Subjects receive 6 month vigorous exercise and subsequent 6 month moderate exercise
  Interventions: Behavioral: Vigorous intensity exercise

INTERVENTIONS:
Behavioral: Non-exercise control — 12 month lifestyle education
  Groups: Non exercise program
Behavioral: Moderate intensity exercise — 12 month moderate intensity exercise by brisk walk 30 min per day and more than 5 days per week.
  Groups: Moderate intensity exercise program
Behavioral: Vigorous intensity exercise — 6 month vigorous intensity exercise on treadmill for 30 min per day and more than 5 days per week, and subsequent 6 month moderate exercise by brisk walk 30 min per day and more than 5 days per week.
  Groups: Vigorous intensity exercise program

SUMMARY:
Our previous randomized controlled trial has recruited 220 subjects with central obesity and allocated the subjects to the non-exercise control, moderate exercise and vigorous exercise groups. The purpose of our previous study was to investigate the effect of moderate and vigorous exercise on improvement of fatty liver. Those subjects will be followed up for incident diabetes at 2 year and 10 year since randomization. The subjects will be invited to participate in on-site visit at 2 and 10 year. Questionaire forms will be collected and fasting plasma glucose level and HbA1c were measured. The history of diabetes and anti-diabetic medication will be recorded. The incident diabetes will be evaluated.

DETAILED DESCRIPTION:
Our previous randomized controlled trial has recruited 220 subject with central obesity and NAFLD. Those subjects were allocated into non-exercise control, moderate exercise and vigorous exercise groups, who received lifestyle education alone, moderate intensity exercise and vigorous intensity exercise, respectively. The exercise intervention lasted one year. Those three group subjects will be followed up and evaluated for incident diabetes at 2 year and 10 year since randomization. All the subjects will be invited to participate in on-site visit at 2 and 10 year. Questionaire forms will be collected and fasting plasma glucose level and HbA1c were measured. The history of diabetes and anti-diabetic medication will be recorded. The incident diabetes will be evaluated.

ELIGIBILITY:
Inclusion criteria

1. Subjects with NAFLD determined by 1H MRS (intrahepatic triglyceride content ≥5%);
2. 40-65 years old;
3. Waist circumference >90cm for men and >85cm for women

Exclusion criteria

1. Consumed more than an average of 140 grams of ethanol (10 alcoholic drinks) per week in men and 70 grams of ethanol (five drinks) in women during the past six months;
2. A history of acute or chronic viral hepatitis, drug-induced liver diseases, and autoimmune hepatitis;
3. Myocardial infarction in the past six months;
4. Biliary obstructive diseases;
5. Uncontrolled hypertension (i.e. systolic BP>180 mmHg, and/or diastolic DBP >100 mmHg);
6. Chronic kidney disease (serum creatinine ≥1.5 mg/dL in men and ≥1.3 mg/dL in women);
7. Heart failure (New York Heart Association III or IV);
8. Currently participating in weight loss programs;
9. Currently pregnant or planning to be pregnant;
10. Having any medical condition that would affect metabolism (i.e. diabetes, known hyperthyroidism or hypothyroidism);
11. Having a medical condition that would limit exercise participation and taking medication that would affect metabolism or weight loss (i.e. thyroid medication and glucocorticoids) or would alter the heart rate response during exercise (i.e. β-blockers);
12. Unable to participate in the follow-up examination.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants in our study included all subjects who had been enrolled in the previous randomized controlled trial.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of type 2 diabetes | 10 years since randomization
  The occurrence of diabetes at 2- and 10-year follow-up

SECONDARY OUTCOMES:
Body weight change | 10 years since randomization
  Body weight change at 2 and 10 year follow-up
Blood pressure change | 10 years since randomization
  Systolic and diastolic blood pressure at 2- and 10-year follow-up
Serum lipid change | 10 years since randomization
  Serum triglyceride, LDL-c levels at 2- and 10- year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: Yes
deidentified data will be available after approval of the proposal
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2023-01~2025-01

REFERENCES:
- [Result] Zhang HJ, He J, Pan LL, Ma ZM, Han CK, Chen CS, Chen Z, Han HW, Chen S, Sun Q, Zhang JF, Li ZB, Yang SY, Li XJ, Li XY. Effects of Moderate and Vigorous Exercise on Nonalcoholic Fatty Liver Disease: A Randomized Clinical Trial. JAMA Intern Med. 2016 Aug 1;176(8):1074-82. doi: 10.1001/jamainternmed.2016.3202. PMID 27379904
- [Result] Zhang HJ, Pan LL, Ma ZM, Chen Z, Huang ZF, Sun Q, Lu Y, Han CK, Lin MZ, Li XJ, Yang SY, Li XY. Long-term effect of exercise on improving fatty liver and cardiovascular risk factors in obese adults: A 1-year follow-up study. Diabetes Obes Metab. 2017 Feb;19(2):284-289. doi: 10.1111/dom.12809. Epub 2016 Nov 22. PMID 27761987
- [Result] Zhang HJ, Zhang XF, Ma ZM, Pan LL, Chen Z, Han HW, Han CK, Zhuang XJ, Lu Y, Li XJ, Yang SY, Li XY. Irisin is inversely associated with intrahepatic triglyceride contents in obese adults. J Hepatol. 2013 Sep;59(3):557-62. doi: 10.1016/j.jhep.2013.04.030. Epub 2013 May 9. PMID 23665283
- [Derived] Chen Y, Chen Z, Pan L, Ma ZM, Zhang H, Li XJ, Li X. Effect of Moderate and Vigorous Aerobic Exercise on Incident Diabetes in Adults With Obesity: A 10-Year Follow-up of a Randomized Clinical Trial. JAMA Intern Med. 2023 Mar 1;183(3):272-275. doi: 10.1001/jamainternmed.2022.6291. PMID 36716009